CLINICAL TRIAL: NCT02339558
Title: Multicenter Phase II Study of Nivolumab in Previously Treated Patients With Recurrent and Metastatic Nasopharyngeal Carcinoma
Brief Title: Nivolumab in Treating Patients With Recurrent and/or Metastatic Nasopharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02673; NCI-2014-02673 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1471; 9742 (Other: Mayo Clinic Cancer Center P2C); 9742 (Other: CTEP); N01CM00099 (NIH); UM1CA186644 (NIH); UM1CA186686 (NIH); UM1CA186691 (NIH)
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Nasopharyngeal Nonkeratinizing Carcinoma; Recurrent Nasopharynx Carcinoma; Stage III Nasopharyngeal Carcinoma AJCC v7; Stage IV Nasopharyngeal Carcinoma AJCC v7; Stage IVA Nasopharyngeal Carcinoma AJCC v7; Stage IVB Nasopharyngeal Carcinoma AJCC v7; Stage IVC Nasopharyngeal Carcinoma AJCC v7
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over approximately 60 minutes on days 1 and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies how well nivolumab works in treating patients with nasopharyngeal cancer that has returned after a period of improvement (recurrent) and/or has spread to other parts of the body (metastatic). Monoclonal antibodies, such as nivolumab, may block tumor growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Objective tumor response to nivolumab in patients with previously treated recurrent and/or metastatic nasopharyngeal carcinoma (NPC) based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.

SECONDARY OBJECTIVES:

I. Tumor response to nivolumab based on immune-related response criteria (IRC). II. Duration of response. III. Progression-free survival and overall survival. IV. Safety and tolerability.

TERTIARY OBJECTIVES:

I. To investigate the effect of nivolumab on tumor burden by analyzing the clearance of plasma Epstein-Barr virus (EBV) deoxyribonucleic acid (DNA) during the first 4-6 weeks of treatment.

II. To investigate the association between treatment outcome and immunological markers: a) Intratumoral expression of programmed cell death 1 (PD-1) and programmed cell death-ligand (PD-L1) in archived NPC tissues (mandatory); b) Serum absolute lymphocyte count at baseline and post-treatment (mandatory); and c) Plasma cytokine levels at baseline and serially during the first 8 weeks of treatment; d) Expression of PD-1 in cluster of differentiation (CD)8+ T cells in tumor infiltrating lymphocytes (TIL) at baseline (optional).

III. To investigate functional magnetic resonance imaging (MRI) sequences as an early predictor of response to nivolumab (optional only at Chinese University of Hong Kong [CUHK]).

OUTLINE:

Patients receive nivolumab intravenously (IV) over approximately 60 minutes on days 1 and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Histologically or cytologically confirmed non-keratinizing nasopharyngeal carcinoma (NPC) that has recurred at locoregional and/or distant sites; NOTE: patients with local recurrence at the bony skull-base as the only site of index disease are excluded; patients with locoregional recurrence without distant metastases must have undergone radical radiotherapy previously
* Measurable disease according to the RECIST criteria (version 1.1), for the evaluation of measurable disease
* Received one or more lines of chemotherapy, which must include prior treatment with a platinum agent and must not be amenable to potentially curative radiotherapy or surgery
* Archived or fresh tumor sample available; willingness to donate blood and tissue for mandatory correlative research studies
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelet count >= 100 x 10^9/L
* Hemoglobin >= 8.0 g/dL
* Serum alanine aminotransferase ([ALT]; serum glutamate-pyruvate transferase [SGPT]), or serum aspartate aminotransferase [AST] where available at the center) < 2.5 x upper limit of normal (ULN), OR < 5 x ULN in the presence of liver metastases
* Serum total bilirubin < 2 x ULN (except patients with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL)
* Serum creatinine < 1.5 x ULN

Exclusion Criteria:

* Any of the following:

  * Chemotherapy =< 4 weeks prior to registration
  * Radiotherapy =< 4 weeks prior to registration
  * Nitrosoureas =< 6 weeks prior to registration or
  * Mitomycin C =< 6 weeks prior to registration
  * Those who have not recovered from adverse events (to grade =< 1 in severity) due to agents administered more than 4 weeks earlier; prior palliative radiotherapy to bone metastases =< 2 weeks prior to registration (i.e. prior palliative radiotherapy to bone metastases is allowed if it is performed > 2 weeks prior to registration)
* Prior investigational agents =< 4 weeks prior to registration
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Known brain metastases or leptomeningeal metastases; NOTE: symptomatic, and/or if they require immunosuppressive doses of corticosteroids (e.g. > 10 mg/day prednisone or equivalents) for at least 2 weeks prior to study drug administration; patients with treated brain metastases who are deemed clinically stable and without radiological progression on positron emission tomography (PET), MRI or computed tomography (CT) scan performed =< 8 weeks of study entry, are not excluded; NOTE: primary nasopharyngeal cancers that directly invade the skull base and extend into the infratemporal fossa (e) are not regarded as brain metastases and are not excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab
* History of severe hypersensitivity reaction to any monoclonal antibody
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception NOTE: breastfeeding should be discontinued if the mother is treated with nivolumab; women of childbearing potential and men must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; they must adhere to contraception for a period of 31 weeks after the last dose of nivolumab
* For patients with unknown human immunodeficiency virus (HIV) status at the time of enrollment, HIV serology must be tested during screening; patients who are tested positive for HIV could be included if there is an adequate cluster of differentiation 4 (CD4) count (> 350/ul) on a stable regimen of highly active anti-retroviral therapy (HAART) with no detectable or minimal viral burden, and no active infections
* For patients with unknown hepatitis B virus surface antigen (HbsAg) status, must be tested during study screening; patients who are tested positive test for HBsAg are excluded if they have inadequately controlled hepatitis B and/or Child-Pugh Class B or C cirrhosis; however, patients with adequately controlled hepatitis are not excluded from the study if they satisfy all of the following criteria: (i) must be receiving a nucleoside analog anti-viral drug for 3 or more months; and (ii) have a serum hepatitis B virus (HBV) deoxyribonucleic acid (DNA) level of less than 100 IU/ml via polymerase chain reaction quantification assays prior to enrollment
* For patients with unknown hepatitis C virus ribonucleic acid (HCV antibody) status, must be tested during study screening; patients who are tested positive for HCV antibody are excluded from the study if they have inadequately controlled hepatitis C and/or Child-Pugh Class B or C cirrhosis; patients with adequately controlled hepatitis are not excluded from the study as defined by having undetectable level of serum HCV antibody level prior to enrollment; patients who are currently on interferon or other anti-HCV therapy will be excluded from study
* Active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids; NOTE: these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded; patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if =< 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Evidence of active or acute (i.e. current, or recent within 4 weeks prior to registration) diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation; patients with abdominal carcinomatosis, a history of non-recent intra-abdominal abscess, or a history of non-recent GI obstruction should be evaluated for the potential need for additional treatment before coming on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2018-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigette B Ma, Principal Investigator — Mayo Clinic Cancer Center P2C
Locations (19):
- United States (15):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Mayo Clinic Cancer Center P2C, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
- Chinese University of Hong Kong-Prince of Wales Hospital, Shatin, Hong Kong, China
- Singapore (3):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre, Singapore
  - Johns Hopkins Singapore, Singapore

REFERENCES:
- [Derived] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Nivolumab): Patients receive 3 mg/kg nivolumab IV over approximately 60 minutes on days 1 and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Nivolumab)
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients that registered for protocol treatment are included in this analysis.
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 57 [37 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 37
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  Singapore | 21
  United States | 16
  China | 8

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response Rate (Complete Response or Partial Response) Based on RECIST Version 1.1
Description: Confirmed response rate is defined as either a Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1. > To be consider a CR, there must be a disappearance of all target lesions and each target lymph node must have reduction in short axis to < 1.0 cm.> > To be considered a PR, at least a 30% decrease in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the baseline value.>
  > The confirmed response rate is reported as the number of patients reporting a CR or PR divided by the total number of evaluable patients multiplied by 100 (reported as a percentage).
Time Frame: Up to 3 years
Population: One patient was a protocol violation and was not included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients with a response
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 44
percentage of patients with a response | 20.5 [9.8 to 35.3]

2. Secondary Outcome: Adverse Events
Description: Adverse events were collected and recorded according to the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine adverse event patterns. For this outcome measure, we summarize the worst graded adverse event regardless of treatment attribution per patient. All reported adverse events are reported in the Adverse Events section of this report.
Time Frame: Up to 3 years on treatment
Population: All patients that began protocol treatment are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 45
Participants
  Grade 3 or higher | 28
  Grade 4 or higher | 5
  Grade 5 | 3

3. Secondary Outcome: Tumor Response to Nivolumab Based on the Immune Response Criteria (IRC)
Description: The Immune Response Criteria (IRC) is a response criteria derived from the WHO criteria.
Time Frame: Up to 3 years
Population: Data was not collected to analyze this secondary endpoint.
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response
Description: Duration of response defined as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented, assessed according to RECIST version 1.1.
Time Frame: Up to 3 years
Population: All patients that reported a CR or PR on treatment were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 9
months | 9.3 [3.6 to 13.1]

5. Secondary Outcome: Progression-free Survival (PFS) Based on RECIST Version 1.1
Description: Progression Free Survival is defined as the time from registration to the time of death or progression, whichever occurs first. The distribution of PFS will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to the first of either death due to any cause or progression, assessed up to 3 years
Population: One patient was ineligible for this endpoint due to a protocol violation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 44
months | 2.8 [1.8 to 7.4]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from registration to the time of death. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to death due to any cause, assessed up to 3 years
Population: One patient was ineligible for this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 44
months | 17.1 [10.9 to NA] — Too few events were recorded to estimate the upper 95% confidence interval.

7. Other Pre Specified Outcome: Clearance of EBV DNA
Description: Plasma EBV DNA half-life during the first 6 weeks of treatment will be correlated with RECIST-response to nivolumab.
Time Frame: Up to 6 weeks of treatment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Intratumoral Expression of PD-1 and PD-L1
Description: PD-1 and PD-L1 expression will be associated with treatment outcomes. The Chi-Square (or Fisher's Exact test) will be used to assess the association of categorical clinical data with categorical biomarker data. Time-to-event clinical data (PFS, OS) will be correlated with biomarker data using Kaplan-Meier methodology and Cox regression models. Logistic regression models will also be used to predict binary clinical data with baseline biomarker data. Finally, graphical methods and descriptive statistics will be used to summarize the data as well.
Time Frame: Baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Serum Absolute Lymphocyte Count
Description: The Chi-Square (or Fisher's Exact test) will be used to assess the association of categorical clinical data with categorical biomarker data. Time-to-event clinical data (PFS, OS) will be correlated with biomarker data using Kaplan-Meier methodology and Cox regression models. Logistic regression models will also be used to predict binary clinical data with baseline biomarker data. Finally, graphical methods and descriptive statistics will be used to summarize the data as well.
Time Frame: Baseline and up to 3 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Expression of PD-1 in CD8+ T Cells in TIL
Description: as for outcome 9
Time Frame: Baseline
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Functional MRI Parameters
Description: Graphical methods and descriptive statistics will be used.
Time Frame: Up to 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were recorded after every 28 day cycle, up to 42 cycles.
Description: Adverse events were recorded after every 28 day cycle, up to 42 cycles.
Arm/Group | Treatment (Nivolumab)
All-Cause Mortality (participants affected / at risk) | 3/45
Serious Adverse Events (participants affected / at risk) | 21/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab) (N=45)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Papilledema (Eye disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 3 (4)
Sepsis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab) (N=45)
Anemia (Blood and lymphatic system disorders) | 8 (22)
Hemolysis (Blood and lymphatic system disorders) | 1 (2)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (4)
Sinus tachycardia (Cardiac disorders) | 1 (12)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (3)
Ear pain (Ear and labyrinth disorders) | 2 (6)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (10)
Endocrine disorders - Other, specify (Endocrine disorders) | 2 (3)
Hyperthyroidism (Endocrine disorders) | 1 (3)
Hypothyroidism (Endocrine disorders) | 8 (26)
Blurred vision (Eye disorders) | 2 (7)
Conjunctivitis (Eye disorders) | 1 (3)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Floaters (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (13)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (9)
Constipation (Gastrointestinal disorders) | 4 (20)
Diarrhea (Gastrointestinal disorders) | 7 (13)
Dry mouth (Gastrointestinal disorders) | 5 (21)
Dysphagia (Gastrointestinal disorders) | 2 (10)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (11)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 7 (8)
Chills (General disorders) | 4 (5)
Edema face (General disorders) | 2 (2)
Edema limbs (General disorders) | 2 (4)
Fatigue (General disorders) | 21 (79)
Fever (General disorders) | 5 (8)
Flu like symptoms (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (6)
Non-cardiac chest pain (General disorders) | 3 (3)
Pain (General disorders) | 9 (18)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 2 (7)
Lung infection (Infections and infestations) | 1 (2)
Paronychia (Infections and infestations) | 1 (2)
Rash pustular (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (5)
Fall (Injury, poisoning and procedural complications) | 1 (3)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (10)
Alkaline phosphatase increased (Investigations) | 3 (8)
Aspartate aminotransferase increased (Investigations) | 7 (22)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 4 (10)
Investigations - Other, specify (Investigations) | 3 (3)
Lipase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 6 (23)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Serum amylase increased (Investigations) | 3 (9)
Weight gain (Investigations) | 1 (16)
Weight loss (Investigations) | 6 (16)
White blood cell decreased (Investigations) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 8 (21)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (31)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 6 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (8)
Hyponatremia (Metabolism and nutrition disorders) | 11 (27)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (11)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (8)
Headache (Nervous system disorders) | 2 (5)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (2)
Paresthesia (Nervous system disorders) | 2 (4)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (10)
Anxiety (Psychiatric disorders) | 2 (4)
Confusion (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (10)
Urinary incontinence (Renal and urinary disorders) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (12)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (21)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (18)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (6)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 3 (33)
Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT02339558/Prot_SAP_000.pdf